CLINICAL TRIAL: NCT02342158
Title: Identifying Molecular Alterations to Guide Individualized Treatment in Advanced Solid Tumors-PERMED01-IPC 2014-003
Brief Title: Identifying Molecular Alterations to Guide Individualized Treatment in Advanced Solid Tumors
Acronym: PERMED01
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institut Paoli-Calmettes (Other)
Collaborators: Cancer Research Center of Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PERMED01-IPC 2014-003
Record Dates: First submitted 2014-12-16; First posted 2015-01-19 (Estimated); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Neoplasm Metastasis
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Biopsy; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Locally advanced /metastatic cancer (Experimental)
  Interventions: Procedure: biopsy or surgical sampling; Other: blood sampling

INTERVENTIONS:
Procedure: biopsy or surgical sampling
Other: blood sampling

SUMMARY:
PERMED01 is a prospective monocenter clinical trial which aims to evaluate the number patients with locally advanced or metastatic cancer for whom identification of molecular alterations in tumor samples can lead to the delivery of a targeted therapy. PERMED01 will enroll 460 patients in 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years
* Histological diagnosis of cancer
* Locally advanced or metastatic, biopsiable disease
* ECOG Performans Status ≤2
* Affiliation to social security
* Signed informed consent.

Exclusion Criteria:

* Emergency, Individually deprived of liberty or placed under the authority of a tutor
* Patients with symptomatic or progressive brain metastasis
* Patients who have only bone and/or brain metastases
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Actual)
Dates: Start 2014-11-12 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
proportion of screened patients in whom a molecular abnormality for which a targeted therapy exists | 4-6 weeks after biopsy

SECONDARY OUTCOMES:
Molecular Characterization of locally advanced and metastatic malignancies using next generation sequencing | 3.5 years
Full exome and transcriptome sequencingof locally advanced and metastatic tumours | 6 years
Circulating tumor DNA detection and characterization in locally advanced and metastatic disease | 4 years
Circulating Tumor Cells (CTC) detection and characterization in breast cancer | 3.5 years
  Comparison of three distinct methods for the CTC detection in blood
Preclinical predictive clinical models validation (limited to breast cancer) | 4 years
  Patient-derived tumour xenograft models (PDX), drug sensitivity tests in vitro

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Paoli-Calmettes, Marseille, France

REFERENCES:
- [Derived] Sabatier R, Garnier S, Guille A, Carbuccia N, Pakradouni J, Adelaide J, Provansal M, Cappiello M, Rousseau F, Chaffanet M, Birnbaum D, Mamessier E, Goncalves A, Bertucci F. Whole-genome/exome analysis of circulating tumor DNA and comparison to tumor genomics from patients with heavily pre-treated ovarian cancer: subset analysis of the PERMED-01 trial. Front Oncol. 2022 Jul 29;12:946257. doi: 10.3389/fonc.2022.946257. eCollection 2022. PMID 35965534
- [Derived] Bertucci F, Goncalves A, Guille A, Adelaide J, Garnier S, Carbuccia N, Billon E, Finetti P, Sfumato P, Monneur A, Pecheux C, Khran M, Brunelle S, Mescam L, Thomassin-Piana J, Poizat F, Charafe-Jauffret E, Turrini O, Lambaudie E, Provansal M, Extra JM, Madroszyk A, Gilabert M, Sabatier R, Vicier C, Mamessier E, Chabannon C, Pakradouni J, Viens P, Andre F, Gravis G, Popovici C, Birnbaum D, Chaffanet M. Prospective high-throughput genome profiling of advanced cancers: results of the PERMED-01 clinical trial. Genome Med. 2021 May 18;13(1):87. doi: 10.1186/s13073-021-00897-9. PMID 34006291